CLINICAL TRIAL: NCT00882700
Title: A Single Center, Open, Randomized, 2-Way, 2-Period, 2-Sequence Crossover Study of the Bioequivalence of 300 mg Cefdinir (Test Formulation) and Omnicel 300 mg Capsule (Reference Formulation) Each Given as a Single Oral Dose to Twenty-Eight Healthy Male and/or Female Volunteers in the Fasting State
Brief Title: To Demonstrate the Relative Bioequivalence of Cefdinir and Omnicef 300 mg Capsule Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 50038
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-04

CONDITIONS: Healthy
Keywords: Antibiotic
MeSH Terms: interventions — Cefdinir

ARMS (2):
- 1 (Experimental): Cefdinir 300 mg Capsule (Sandoz, Austria)
  Interventions: Drug: Cefdinir 300 mg Capsule (Sandoz, Austria)
- 2 (Active Comparator): Omnicef Cefdinir 300 mg Capsule (Abbott Laboratories, USA)
  Interventions: Drug: Omnicef Cefdinir 300 mg Capsule (Abbott Laboratories, USA)

INTERVENTIONS:
Drug: Cefdinir 300 mg Capsule (Sandoz, Austria)
  Arms: 1
Drug: Omnicef Cefdinir 300 mg Capsule (Abbott Laboratories, USA)
  Arms: 2

SUMMARY:
To demonstrate the relative bioequivalence of Cefdinir and Omnicel 300 mg capsule fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2005-04; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, M.D., Principal Investigator — SFBC Anapharm